CLINICAL TRIAL: NCT00567606
Title: Prevention of Osteoporosis in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0536-01-FB; 1R01NR007743-04 (NIH)
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength/Weight Training (Experimental): Subjects in the G1 group receive drug/supplement combination and strength/weight training exercises for upper and lower extremities and the spine.
  Interventions: Other: Strength/Weight Training & Drug/Supplement
- Drug Supplement only (Experimental): Subjects in the G2 group receive drug/supplement combination, but do not participate in strength/weight training exercises.
  Interventions: Combination Product: Drug/Supplement only

INTERVENTIONS:
Other: Strength/Weight Training & Drug/Supplement — G1 group receives 1200 mg of calcium and 400 IU of vitamin D supplements per day, 35 mg of risedronate per week and strength/weight training exercises for upper and lower extremities and the spine.
  Other Names: Actonel
  Arms: Strength/Weight Training
Combination Product: Drug/Supplement only — G2 group receives 1200 mg of calcium and 400 IU of vitamin D supplements per day, 35 mg of risedronate per week, but do not participate in strength/weight training exercises.
  Other Names: Actonel
  Arms: Drug Supplement only

SUMMARY:
The purpose of this study is to test whether strength/weight training exercises enhance the effectiveness of calcium, vitamin D, and risedronate for the prevention and treatment of osteoporosis in postmenopausal breast cancer survivors.

DETAILED DESCRIPTION:
Each year, more than 192,200 women are diagnosed with breast cancer (Greenlee, Hill-Harmon, Murray, & Thun, 2001). With an increase in early detection and improved therapies, more of these women have become survivors (Vassilopoulou-Sellin & Theriault, 1994). However, many of these women are at increased risk for osteoporosis and the debilitating consequences. This increased risk occurs for two reasons. Over 50-70% of women under the age of 50 (premenopausal) who are treated with adjuvant chemotherapy experience ovarian failure and early menopause (Ali & Twibel, 1994; Cobleigh et al., 1994; Samaan et al., 1978), resulting in a long postmenopausal period of estrogen deprivation. Breast cancer survivors also are at greater risk for osteoporosis because they usually are not candidates for hormone replacement therapy (HRT). Estrogen can influence the growth of cancer in women, especially those with estrogen receptor positive tumors (ER+), and at least 60% of women have ER+ breast cancer (DeVita, Hellman & Rosenberg, 1997). While the use of HRT significantly reduces osteoporosis and the risk of forearm, vertebral, pelvic, and hip fractures in postmenopausal women (Cobleigh et al., 1994; Finkelstein, 1996), women with a history of breast cancer generally are not considered candidates for HRT. Without estrogen, women may lose up to 30% of their bone mass within the first 5-years postmenopause, with continued bone loss over time, but at a slower rate. Very little information has been reported on the incidence and treatment of osteoporosis in breast cancer survivors (Headley et al., 1998; Hosking et al., 1998).

Osteoporosis is a major risk factor for chronic disability and especially hip fractures. The majority of individuals with hip fractures never return to prefracture functional status and estimates of health care costs for individuals with osteoporosis exceed the costs for those with congestive heart failure or with asthma (U.S. Congress Office of Technology Assessment, 1994; Ray, Chan, Thamer & Meltin, 1997). Prevention and treatment of osteoporosis, by increasing bone mineral density (BMD) and muscle strength, may decrease the chronic disabilities associated with osteoporosis and improve quality and quantity of life (Mahon, 1998). Research on effective alternatives to HRT for the prevention of osteoporosis in breast cancer survivors has been targeted as a priority area by the Office of Cancer Survivorship (Division of Cancer Control and Population Sciences) at the National Cancer Institute (Office of Cancer Survivorship, 1999). No reports were found in which the effectiveness of the combination of risedronate, calcium, and vitamin D (administered together and at the current recommended levels for postmenopausal women) was studied, nor has the effectiveness of the addition of long term progressive strength/weight training exercises been evaluated in this at risk population of breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* read, speak and understand English;
* be female;
* be between the ages of 35 and 75;
* have completed treatment (except tamoxifen) for stage 0, I or II breast cancer (i.e. surgery, chemotherapy, radiation) at least 6 months prior to admission to the study;
* be 1 year postmenopausal (12-months amenorrheic; subjects 55-years or younger with history of hysterectomy without oophorectomy must have it confirmed by two baseline measures of FSH >40 IU/ml);
* have a BMD T-score of -1.0 SD or lower at one or more sites (spine, hip or forearm); and
* have agreement of their primary care provider for participation in the study.

Exclusion Criteria:

* have a recurrence of their breast cancer;
* currently take hormone replacement therapy, bisphosphonates, calcitonin, raloxifene, calcitriol, or glucocorticosteroids.;
* currently do strength/weight training exercises or high impact exercises (such as running, jumping rope, high impact aerobic dance, martial arts, volleyball, or basketball) two to three times weekly;
* have a body mass index (BMI) equal to or greater than 35;
* have serum calcium, creatinine or TSH (if on thyroid therapy) outside the normal limits;
* have active gastrointestinal problems such as dysphagia, esophageal disease, gastritis, duodenitis, or ulcers;
* have Paget=s disease;
* have renal disease (renal stones or serum creatinine levels greater than the upper normal limits);
* have a recent history of a spinal fracture (within the past 6 months);
* have features of an acute fracture on baseline spinal x-rays;
* have other concomitant conditions that prohibit strength/weight training exercises, calcium, or vitamin D intake.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2002-04-01 (Actual); Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | at 12, 24, and 36 months
  Bone Mineral Density (gm/cm2) will be measured by Dual-Energy X-ray Absorptiometry (DEXA) of the hip, spine and forearm

SECONDARY OUTCOMES:
Muscle Strength | at baseline, 6, 12, 24, and 36 months
  Muscle Strength (peak torque/body weight at 60 degrees) will be assessed using BiodexTM Velocity Spectrum Evaluation (Medical Systems, Inc., 1993)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Waltman, PhD, ARNP, Principal Investigator — University of Nebraska Medical Center, College of Nursing
Locations (4):
- United States (4):
  - University of Nebraska Medical Center, College of Nursing, Kearney, Nebraska
  - University of Nebraska Medical Center, College of Nursing, Lincoln, Nebraska
  - University of Nebraska Medical Center, College of Nursing, Omaha, Nebraska
  - University of Nebraska Medical Center, College of Nursing, Scottsbluff, Nebraska

REFERENCES:
- [Result] Twiss JJ, Gross GJ, Waltman NL, Ott CD, Lindsey AM. Health behaviors in breast cancer survivors experiencing bone loss. J Am Acad Nurse Pract. 2006 Oct;18(10):471-81. doi: 10.1111/j.1745-7599.2006.00165.x. PMID 16999712
- [Result] Ott CD, Twiss JJ, Waltman NL, Gross GJ, Lindsey AM. Challenges of recruitment of breast cancer survivors to a randomized clinical trial for osteoporosis prevention. Cancer Nurs. 2006 Jan-Feb;29(1):21-31, quiz 32-3. doi: 10.1097/00002820-200601000-00004. PMID 16557117